CLINICAL TRIAL: NCT04488393
Title: Clinical Performance of NIPT (Noninvasive Prenatal Testing) in Multiple Gestation Pregnancies (SCMM-T21-110)
Brief Title: Clinical Performance of NIPT in Multiple Gestation Pregnancies
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: Sequenom, Inc/Laboratory Corporation of America Holdings (Unknown)
Responsible Party: Principal Investigator, Lorraine Dugoff, Professor of Obstetrics and Gynecology, University of Pennsylvania
Other Study IDs: SCMM-T21-110
Record Dates: First submitted 2020-07-22; First posted 2020-07-28 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2022-12

CONDITIONS: Trisomy 21 in Fetus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pregnancies with multiple gestations
  Interventions: Device: MaterniT21 PLUS and GENOME Laboratory-Developed Tests

INTERVENTIONS:
Device: MaterniT21 PLUS and GENOME Laboratory-Developed Tests — Both the MaterniT21 PLUS and GENOME are intended for use as laboratory developed test that analyze ccfDNA extracted from a maternal blood sample utilizing Massively Parallel Sequencing (MPS) technology.

SUMMARY:
This study plans to evaluate the clinical performance of the MaterniT21 PLUS and/or GENOME Laboratory Developed Test, in the detection of fetal trisomy 21 in circulating cell-free DNA extracted from maternal blood samples obtained from women pregnant with a twin gestation.

ELIGIBILITY:
Inclusion Criteria:

* subject pregnant with a multiple gestation and received NIPT from Sequenom Laboratories;
* subject was 18 or older at the time of NIPT

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: The Study Population will consist of women 18 years of age and older who underwent testing with a Sequenom NIPT, were pregnant with a multiple gestation at the time of testing and whose pregnancies should have outcome based upon gestational age at the time of testing.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-11-15 (Actual); Study Completion 2022-06-19 (Actual)

PRIMARY OUTCOMES:
Determination of sensitivity of NIPT detection of trisomy 21 among a population of women with twin gestations. | time from maternal blood draw to delivery
Determination of specificity of NIPT detection of trisomy 21 among a population of women with twin gestations. | time from maternal blood draw to delivery

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Siegel MR, James K, Bromley B, Koelper NC, Chasen ST, Griffin L, Roman AS, Limaye M, Ranzini A, Clifford C, Biggio JR, Subramaniam A, Seasely AR, Page JM, Nicholas SS, Idler J, Rao R, Shree R, McLennan G, Dugoff L; Twin cfDNA Study Consortium. First-Trimester Cell-Free DNA Fetal Fraction and Birth Weight in Twin Pregnancies. Am J Perinatol. 2025 Apr;42(5):605-611. doi: 10.1055/a-2413-2353. Epub 2024 Sep 11. PMID 39260415